CLINICAL TRIAL: NCT01978184
Title: Randomized Phase II Trial of Pre-Operative Gemcitabine and Nab Paclitacel With or With Out Hydroxychloroquine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nathan Bahary, MD (Other)
Responsible Party: Sponsor-Investigator, Nathan Bahary, MD, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCI# 13-074
Record Dates: First submitted 2013-10-30; First posted 2013-11-07 (Estimated); Results first posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer, resectable adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Albumin-Bound Paclitaxel; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gemcitabine and abraxane (Experimental): Gemcitabine and Abraxane will be administered on an outpatient basis on Days 3, 10, 17, 31, 38, and 45 as an intravenous infusion. The dose on Day 3 will be 1000 mg/m of gemcitabine followed by a 125 mg/m2 of abraxane and the infusion will take 1 hour. The second dose and infusion time may be decreased. Prior to each gemcitabine infusion, subjects will be pre-medicated with an FDA-approved anti-emetic (anti-nausea medication) in an effort to prevent nausea, at the discretion of the study physician.
  Interventions: Drug: gemcitabine; Drug: abraxane
- gemcitabine, abraxane and hydroxychloroquine (Experimental): Gemcitabine and Abraxane will be administered on an outpatient basis on Days 3, 10, 17, 31, 38, and 45 as an intravenous infusion. The dose on Day 3 will be 1000 mg/m of gemcitabine followed by a 125 mg/m2 of abraxane and the infusion will take 1 hour. The second dose and infusion time may be decreased. Prior to each gemcitabine infusion, subjects will be pre-medicated with an FDA-approved anti-emetic (anti-nausea medication) in an effort to prevent nausea, at the discretion of the study physician.
  Hydroxychloroquine is an oral drug (capsule) that subjects will take once or twice a day at home. The dose of hydroxychlorquien will be 1200mg. This is an experimental drug. Subjects will take their first dose of hydroxychloroquine on Day 1 (48 hours before the first infusion of gemcitabine/abraxane), and will continue to take it every day until the day before surgery.
  Interventions: Drug: gemcitabine; Drug: abraxane; Drug: hydroxychloroquine

INTERVENTIONS:
Drug: gemcitabine
  Other Names: Gemzar
Drug: abraxane
  Other Names: nab-Paclitacel
Drug: hydroxychloroquine
  Other Names: Plaquenil
  Arms: gemcitabine, abraxane and hydroxychloroquine

SUMMARY:
This is a randomized phase II trial that will examine the ability of the hydroxychloroquine to improve the clinical activity of a pre-operative regimen of gemcitabine and nab-paclitaxel in subjects with potentially resectable adenocarcinoma of the pancreas. Eligible subjects will receive 2 cycles of gemcitabine and nab-paclitaxel (day 1, 8, 15) with or without hydrocychloroquine followed by surgical resection. Primary endpoint will be histologic response as graded by Evans criteria. Secondary endpoints will be CA19-9 response and PET response. Pre and post treatment tissue biopsies will be obtained to assess for levels of autophagy in tumor, liver and peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with biopsy-proven potentially resectable or borderline adenocarcinoma of the pancreas as determined by National Comprehensive Cancer Network (NCCN) criteria
* Karnofsky performance status of 70-100%
* No active second malignancy except for basal cell carcinoma of the skin
* Patient has adequate biological parameters as demonstrated by the following blood counts at screening
* Absolute neutrophil count (ANC) ≥1.5 × 109/L;
* Platelet count ≥100,000/mm3 (100 × 109/L);
* Hemoglobin (Hgb) ≥9 g/dL.
* Patient has the following blood chemistry levels at Baseline
* aspartate aminotransferase (AST) (SGOT), Alanine transaminase (SGPT) ≤2.5 × upper limit of normal range (ULN)
* Total bilirubin ≤ULN
* Serum Creatinine ≤ 1.5mg/dl OR calculated creatinine clearance ≥ 50 for those patients with creatinine greater than 1.5
* Prothrombin time (PT)within normal limits (WNL). If patient is on warfarin for prophylactic clot presentation for indwelling catheter, Partial PT/PTT may be +/- 15 %
* thromboplastin time (PTT) WNL. If patient on warfarin for prophylactic clot presentation for indwelling catheter, PT/PTT may be +/- 15 %
* Age >18 years.
* Patient must be able to swallow enteral medications with no requirement for a feeding tube. Patient's must not have intractable nausea or vomiting which prohibits the patient from oral medications
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Subjects deemed surgically unresectable or subjects unwilling to undergo surgical resection.
* Subjects who have received chemotherapy within 12 months prior to randomization.
* Prior use of radiotherapy or investigational agents for pancreatic cancer.
* Any evidence of metastasis to distant organs (liver, lung, peritoneum).
* Symptomatic evidence of gastric outlet obstruction
* Inability to adhere to study and/or follow-up procedures
* History of allergic reactions or hypersensitivity to the study drugs (hydroxychloroquine, gemcitabine, abraxane).
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. All females of childbearing potential must have a blood test or urine study within two weeks prior to randomization to rule out pregnancy.
* Patients with porphyria are ineligible.
* Patients with psoriasis are ineligible unless the disease is well controlled and they are under the care of a specialist who agrees to monitor the patient for exacerbations.
* Patients requiring the use of enzyme-inducing anti-epileptic medication that includes: phenytoin, carbamazepine, phenobarbital, primidone or oxcarbazepine are excluded.
* Patients with previously documented macular degeneration or diabetic retinopathy are excluded.
* Baseline electrocardiogram (EKG) with corrected QT interval (QTc) >470 msec (including subjects on medication). Subjects with ventricular pacemaker for whom QT interval is not measurable will be eligible on a case-by-case basis.
* Patient with a history of interstitial lung disease, history of slowly progressive dyspnea, sarcoidosis, silicosis, idiopathic pulmonary fibrosis or pulmonary hypersensitivity pneumonitis
* Patient with known active infection with HIV, Hepatitis B or Hepatitis C
* Patients requiring use of warfarin for therapeutic purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-11; Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Zeh, MD, Principal Investigator — University of Pittsburgh CancerCenters
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Miller-Ocuin JL, Liang X, Boone BA, Doerfler WR, Singhi AD, Tang D, Kang R, Lotze MT, Zeh HJ 3rd. DNA released from neutrophil extracellular traps (NETs) activates pancreatic stellate cells and enhances pancreatic tumor growth. Oncoimmunology. 2019 Jun 11;8(9):e1605822. doi: 10.1080/2162402X.2019.1605822. eCollection 2019. PMID 31428515
- [Derived] Boone BA, Murthy P, Miller-Ocuin J, Doerfler WR, Ellis JT, Liang X, Ross MA, Wallace CT, Sperry JL, Lotze MT, Neal MD, Zeh HJ 3rd. Chloroquine reduces hypercoagulability in pancreatic cancer through inhibition of neutrophil extracellular traps. BMC Cancer. 2018 Jun 22;18(1):678. doi: 10.1186/s12885-018-4584-2. PMID 29929491

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine + Abraxane: Gemcitabine and Abraxane administered as an intravenous infusion on Study Days 3, 10, 17, 31, 38, and 45. Day 3 dosing: 1 hour infusion - 1000 mg/m^2 of gemcitabine followed by a 125 mg/m^2 of abraxane. Prior to each gemcitabine infusion, subjects were pre-medicated with an FDA-approved anti-emetic (anti-nausea medication) in an effort to prevent nausea, at the discretion of the study physician.
- Gemcitabine + Abraxane and Hydroxychloroquine: Gemcitabine and Abraxane administered as an intravenous infusion on Study Days 3, 10, 17, 31, 38, and 45. Day 3 dosing: 1 hour infusion - 1000 mg/m^2 of gemcitabine followed by a 125 mg/m^2 of abraxane. Prior to each gemcitabine infusion, subjects were pre-medicated with an FDA-approved anti-emetic (anti-nausea medication) in an effort to prevent nausea, at the discretion of the study physician.
  Hydroxychloroquine oral capsules taken once or twice a daily at a dose of 1200mg. The first dose of hydroxychloroquine taken on Day 1 (48 hours before the first infusion of gemcitabine/abraxane), and continued daily until one day before surgery.
Period: Overall Study
Arm/Group | Gemcitabine + Abraxane | Gemcitabine + Abraxane and Hydroxychloroquine
Started | 43 | 61
Completed | 30 | 41
Not Completed | 13 | 20
Not completed — Progressive disease | 5 | 5
Not completed — Other than PDA | 2 | 2
Not completed — Physician Decision | 0 | 3
Not completed — Noncompliance | 1 | 2
Not completed — Death | 1 | 0
Not completed — Withdrew- toxicities or physical decline | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gemcitabine + Abraxane | Gemcitabine + Abraxane and Hydroxychloroquine | Total
Number analyzed (Participants) | 30 | 41 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (11.8) | 66.1 (8.4) | 65 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 31
  Male | 16 | 24 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 30 | 40 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 28 | 38 | 66
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Evans Grade Histopathologic Response
Description: The number of patients who exhibited an Evans grade Histologic response (I, IIA, IIB, or III) to pre-operative gemcitabine / nab-paclitaxel. Histological response validated scoring system by Evans is as follows: Grade I: 1-9% tumor destruction, Grade II: 10 - 90%, Grade III: >90% tumor destruction (Grade IIA = 10-50% of tumor cells destroyed; Grade IIB = 50-90% of tumor cells destroyed), Grade IV: Absence of viable tumor cells.
Time Frame: Up to 4 years
Population: Patients who went to surgery and were evaluable for Evans Grade Histopathologic Response.
Measure: Number; unit: number of participants
Arm/Group | Gemcitabine + Abraxane | Gemcitabine + Abraxane and Hydroxychloroquine
Number analyzed (Participants) | 30 | 41
number of participants
  Evans grade - I | 10 | 7
  Evans grade - IIA | 17 | 12
  Evans grade - IIB | 3 | 13
  Evans grade - III | 0 | 9

2. Primary Outcome: Age at Diagnosis
Description: The mean age of patients at the time of diagnosis of disease (as a variable in the proportional odds logistic regression, secondary analysis of Evans Grade).
Time Frame: Baseline - At the time of diagnosis, prior to treatment
Population: Patients who went to surgery and were evaluable for Evans Grade Histopathologic Response.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Gemcitabine + Abraxane | Gemcitabine + Abraxane and Hydroxychloroquine
Number analyzed (Participants) | 30 | 41
years | 63.6 (11.8) | 66.1 (8.4)

3. Primary Outcome: CT Tumor Size
Description: Tumor size as measured via computerized tomography (CT) scan (as a variable in the proportional odds logistic regression, secondary analysis of Evans Grade).
Time Frame: Baseline - At the time of diagnosis, prior to treatment
Population: Patients who went to surgery and were evaluable for Evans Grade Histopathologic Response.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Gemcitabine + Abraxane | Gemcitabine + Abraxane and Hydroxychloroquine
Number analyzed (Participants) | 29 | 41
centimeters | 2.562069 (1.105962) | 2.543056 (1.139370)

4. Primary Outcome: Cancer Diagnosis Stage
Description: The number of participants in cancer diagnosis stage groups. Stage 0: cancer hasn't spread to nearby tissues/located in the same of origin.Stage I: cancers hasn't grown deeply into nearby tissues or spread to lymph nodes or other parts of the body. Stage II and III: cancers have grown more deeply into nearby tissues (may have metastasized to lymph nodes but not other parts of the body). Stage IV: most advanced stage (metastatic cancer) ; cancer has spread to other parts of the body. Stages subdivided further into the categories "A" (less agressive disease) and "B" (more advanced cancer). Example: stage IIA is less aggressive than stage IIB, but stage IIIA is more aggressive than stage IIB. (Stage variable used in the proportional odds logistic regression, secondary analysis of Evans Grade).
Time Frame: Baseline - At the time of diagnosis, prior to treatment
Population: Patients who went to surgery and were evaluable for Evans Grade Histopathologic Response.
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine + Abraxane | Gemcitabine + Abraxane and Hydroxychloroquine
Number analyzed (Participants) | 30 | 41
Participants
  IA | 0 | 2
  IB | 5 | 1
  IIA | 6 | 11
  IIB | 19 | 20
  Not Available | 0 | 7

5. Primary Outcome: Type of Surgical Procedure (Operation)
Description: The number of participants in having each type of surgical resection procedure: Celiac Axis Resection With Distal Pancreatectomy (DPCAR) (Modified Appleby), Distal Pancreatectomy, Total Pancreatectomy, or Whipple. (Operation variable used in the proportional odds logistic regression, secondary analysis of Evans Grade).
Time Frame: At the time of surgery (≥2 weeks and ≤6 weeks post chemotherapy)
Population: Patients who went to surgery and were evaluable for Evans Grade Histopathologic Response.
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine + Abraxane | Gemcitabine + Abraxane and Hydroxychloroquine
Number analyzed (Participants) | 30 | 41
Participants
  DPCAR | 2 | 0
  Distal Pancreatectomy | 3 | 5
  Total Pancreatectomy | 1 | 0
  Whipple | 24 | 36

6. Primary Outcome: Robotic Resection Surgery
Description: The number of participants who had robotic resection surgery. (Robotic surgery variable used in the proportional odds logistic regression, secondary analysis of Evans Grade).
Time Frame: At the time of surgery (≥2 weeks and ≤6 weeks post chemotherapy)
Population: Patients who went to surgery and were evaluable for Evans Grade Histopathologic Response.
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine + Abraxane | Gemcitabine + Abraxane and Hydroxychloroquine
Number analyzed (Participants) | 30 | 41
Participants
  Yes - robotic surgical resection procedure | 8 | 10
  No - not robotic surgical resection procedure | 22 | 31

7. Primary Outcome: Age-Adjusted Charlson Comorbidity Index
Description: The Charlson Comorbidity Index is a method of categorizing comorbidities of patients based on the International Classification of Diseases (ICD) diagnosis codes found in administrative data, such as hospital abstracts data. Each comorbidity category has an associated weight (from 1 to 6), based on the adjusted risk of mortality or resource use, and the sum of all the weights results in a single comorbidity score for a patient. A score of zero indicates that no comorbidities were found. The higher the score, the more likely the predicted outcome will result in mortality or higher resource use. Up to 12 comorbidities with various weightings can result in a maximum score of 24. The minimum score is zero.
Time Frame: Prior to treatment
Population: Patients who went to surgery and were evaluable for Evans Grade Histopathologic Response.
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine + Abraxane | Gemcitabine + Abraxane and Hydroxychloroquine
Number analyzed (Participants) | 30 | 41
Participants
  Age-Adjusted CCI=2 | 3 | 1
  Age-Adjusted CCI=3 | 5 | 2
  Age-Adjusted CCI=4 | 7 | 11
  Age-Adjusted CCI=5 | 8 | 15
  Age-Adjusted CCI=6 | 5 | 8
  Age-Adjusted CCI=7 | 2 | 2
  Age-Adjusted CCI=8 | 0 | 2

8. Secondary Outcome: Carbohydrate Antigen 19-9 (CA19-9) Response
Description: Levels of Carbohydrate antigen 19-9 (CA19-9) response to pre-operative gemcitabine/ nab-paclitaxel measured in the serum (original scale)
Time Frame: Prior to treatment (average 73.3 +/- 9.9 days prior to surgery)
Population: Participants that were assigned to treatment and did not withdraw consent prior to being given drug.
Measure: Mean (Standard Deviation); unit: units per milliliter (U/mL)
Arm/Group | Gemcitabine + Abraxane | Gemcitabine + Abraxane and Hydroxychloroquine
Number analyzed (Participants) | 30 | 41
units per milliliter (U/mL) | 351.820 (839.925) | 1534.633 (3558.1212)

9. Secondary Outcome: Carbohydrate Antigen 19-9 (CA19-9) Response
Description: as for outcome 8
Time Frame: After treatment (50-67 days post treatment/surgery)
Population: Participants that were assigned to treatment and did not withdraw consent prior to being given drug.
Measure: Mean (Standard Deviation); unit: units per milliliter (U/mL)
Arm/Group | Gemcitabine + Abraxane | Gemcitabine + Abraxane and Hydroxychloroquine
Number analyzed (Participants) | 29 | 41
units per milliliter (U/mL) | 319.079 (1338.259) | 1696.710 (9850.273)

10. Secondary Outcome: Positive Lymph Node Involvement
Description: The proportion of participants with positive (disease) lymph nodes involvement.
Time Frame: At the time of surgery (≥2 weeks and ≤6 weeks post chemotherapy)
Population: Participants that were assigned to treatment and did not withdraw consent prior to being given drug.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Gemcitabine + Abraxane | Gemcitabine + Abraxane and Hydroxychloroquine
Number analyzed (Participants) | 30 | 41
proportion of participants | 0.8 [0.614 to 0.923] | 0.561 [0.397 to 0.715]

11. Secondary Outcome: Rate of R0 Resection
Description: The proportion of participants having resection for cure or complete remission, in which the surgical margins are negative for tumor cells. R0 resection indicates a microscopically margin-negative resection, in which no gross or microscopic tumor remains in the primary tumor bed.
Time Frame: At the time of surgery (≥2 weeks and ≤6 weeks post chemotherapy)
Population: Participants that were assigned to treatment and did not withdraw consent prior to being given drug.
Measure: Mean (95% Confidence Interval); unit: proportion of participants
Arm/Group | Gemcitabine + Abraxane | Gemcitabine + Abraxane and Hydroxychloroquine
Number analyzed (Participants) | 30 | 41
proportion of participants | 0.7 [0.506 to 0.853] | 0.829 [0.679 to 0.928]

ADVERSE EVENTS:
Time Frame: Up to 4 years
Arm/Group | Gemcitabine + Abraxane | Gemcitabine + Abraxane and Hydroxychloroquine
All-Cause Mortality (participants affected / at risk) | 28/43 | 34/61
Serious Adverse Events (participants affected / at risk) | 30/43 | 39/61
Other Adverse Events (participants affected / at risk) | 43/43 | 60/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine + Abraxane (N=43) | Gemcitabine + Abraxane and Hydroxychloroquine (N=61)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (3)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (3)
Alanine aminotransferase increased (Investigations) | 1 (2) | 6 (21)
Alkaline phosphatase increased (Investigations) | 1 (2) | 1 (3)
Allergic reaction (Immune system disorders) | 1 (2) | 1 (3)
Anemia (Blood and lymphatic system disorders) | 4 (9) | 3 (9)
Aspartate aminotransferase increased (Investigations) | 2 (4) | 4 (12)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (3)
Blood bilirubin increased (Investigations) | 1 (2) | 1 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Catheter related infection (Infections and infestations) | 1 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 5 (21)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 3 (13)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Edema limbs (General disorders) | 0 (0) | 1 (3)
Fatigue (General disorders) | 2 (4) | 5 (18)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (20) | 2 (6)
Fever (General disorders) | 1 (2) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 2 (6)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (9)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (5) | 0 (0)
Hypertension (Vascular disorders) | 4 (10) | 3 (9)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3) | 6 (24)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (6)
Hypotension (Vascular disorders) | 0 (0) | 2 (9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 3 (6) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Lipase increased (Investigations) | 0 (0) | 1 (3)
Lung infection (Infections and infestations) | 2 (4) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 3 (9)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Multi-organ failure (General disorders) | 1 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 3 (12)
Neutrophil count decreased (Investigations) | 10 (30) | 11 (45)
Pain (General disorders) | 1 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Platelet count decreased (Investigations) | 3 (6) | 1 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 0 (0)
Skin infection (Infections and infestations) | 3 (12) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (3) | 1 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (3)
Ventricular fibrillation (Cardiac disorders) | 1 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 2 (6)
White blood cell decreased (Investigations) | 6 (12) | 10 (39)
Wound infection (Infections and infestations) | 2 (5) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine + Abraxane (N=43) | Gemcitabine + Abraxane and Hydroxychloroquine (N=61)
Abdominal pain (Gastrointestinal disorders) | 5 (10) | 8 (24)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 1 (3)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (6)
Alanine aminotransferase increased (Investigations) | 18 (56) | 32 (147)
Alkaline phosphatase increased (Investigations) | 11 (27) | 23 (105)
Allergic reaction (Immune system disorders) | 1 (4) | 1 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (6) | 10 (39)
Anemia (Blood and lymphatic system disorders) | 36 (151) | 50 (333)
Anorexia (Metabolism and nutrition disorders) | 5 (10) | 12 (39)
Anxiety (Psychiatric disorders) | 4 (8) | 3 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 17 (51) | 36 (135)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (6) | 3 (9)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (3)
Blood bilirubin increased (Investigations) | 3 (8) | 7 (27)
Blurred vision (Eye disorders) | 0 (0) | 2 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
CPK increased (Investigations) | 0 (0) | 1 (3)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (2) | 1 (3)
Catheter related infection (Infections and infestations) | 1 (2) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (3)
Chills (General disorders) | 2 (5) | 4 (13)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (3)
Confusion (Psychiatric disorders) | 1 (2) | 1 (3)
Constipation (Gastrointestinal disorders) | 10 (26) | 13 (42)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 2 (6)
Creatinine increased (Investigations) | 4 (8) | 4 (12)
Dehydration (Metabolism and nutrition disorders) | 4 (9) | 9 (36)
Depression (Psychiatric disorders) | 1 (2) | 2 (6)
Diarrhea (Gastrointestinal disorders) | 11 (27) | 25 (100)
Dizziness (Nervous system disorders) | 1 (3) | 3 (9)
Dry mouth (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (9)
Dysgeusia (Nervous system disorders) | 1 (2) | 2 (9)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 5 (18)
Edema limbs (General disorders) | 8 (18) | 7 (21)
Edema trunk (General disorders) | 1 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 1 (3)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Esophageal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (6)
Fatigue (General disorders) | 29 (86) | 27 (141)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (28) | 7 (27)
Fever (General disorders) | 6 (16) | 8 (28)
Flatulence (Gastrointestinal disorders) | 3 (10) | 5 (15)
Flu like symptoms (General disorders) | 1 (2) | 4 (12)
Flushing (Vascular disorders) | 0 (0) | 1 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (6) | 4 (15)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (4) | 7 (24)
General disorders and administration site conditions - Other, specify (General disorders) | 5 (20) | 7 (24)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 10 (57)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (3)
Headache (Nervous system disorders) | 1 (2) | 3 (9)
Hematoma (Vascular disorders) | 1 (2) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (3)
Hemoglobin increased (Investigations) | 1 (2) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (3)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Hot flashes (Vascular disorders) | 0 (0) | 1 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (3) | 3 (9)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (30) | 3 (9)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (4) | 1 (3)
Hypernatremia (Metabolism and nutrition disorders) | 2 (5) | 2 (6)
Hypertension (Vascular disorders) | 13 (59) | 14 (60)
Hypoalbuminemia (Metabolism and nutrition disorders) | 25 (92) | 40 (204)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (4) | 6 (30)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (2) | 1 (3)
Hypokalemia (Metabolism and nutrition disorders) | 11 (33) | 20 (81)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 3 (9)
Hyponatremia (Metabolism and nutrition disorders) | 17 (53) | 28 (150)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (3) | 4 (24)
Hypotension (Vascular disorders) | 1 (2) | 9 (33)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 3 (8) | 2 (6)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Insomnia (Psychiatric disorders) | 1 (2) | 5 (15)
Investigations - Other, specify (Investigations) | 0 (0) | 3 (9)
Lipase increased (Investigations) | 1 (3) | 1 (3)
Lung infection (Infections and infestations) | 2 (4) | 0 (0)
Lymphocyte count decreased (Investigations) | 13 (37) | 13 (63)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 1 (3)
Malaise (General disorders) | 1 (2) | 3 (9)
Memory impairment (Nervous system disorders) | 1 (2) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2 (10) | 5 (18)
Mucosal infection (Infections and infestations) | 1 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (4) | 2 (6)
Multi-organ failure (General disorders) | 1 (3) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (3)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 (4) | 2 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (3)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (3)
Nausea (Gastrointestinal disorders) | 12 (41) | 31 (126)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (2) | 3 (12)
Neutrophil count decreased (Investigations) | 29 (123) | 41 (198)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (3)
Pain (General disorders) | 5 (15) | 4 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (12)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (6)
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (6) | 6 (24)
Phlebitis (Vascular disorders) | 0 (0) | 1 (3)
Platelet count decreased (Investigations) | 30 (113) | 45 (228)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (6)
Pulmonary valve disease (Cardiac disorders) | 0 (0) | 1 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (9)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (12)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (2) | 1 (3)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (2) | 0 (0)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 (0) | 1 (3)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 6 (18)
Serum amylase increased (Investigations) | 0 (0) | 1 (3)
Sinus bradycardia (Cardiac disorders) | 1 (4) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 2 (6)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (5) | 8 (33)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Skin infection (Infections and infestations) | 3 (20) | 1 (6)
Somnolence (Nervous system disorders) | 0 (0) | 1 (4)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Superficial thrombophlebitis (Vascular disorders) | 0 (0) | 1 (3)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (3)
Thromboembolic event (Vascular disorders) | 1 (5) | 2 (7)
Tooth infection (Infections and infestations) | 0 (0) | 1 (3)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (3)
Tremor (Nervous system disorders) | 0 (0) | 1 (3)
Tricuspid valve disease (Cardiac disorders) | 0 (0) | 1 (3)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (6)
Urinary tract infection (Infections and infestations) | 0 (0) | 5 (18)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (3)
Vascular disorders - Other, specify (Vascular disorders) | 1 (2) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (3) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (3)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (3)
Vomiting (Gastrointestinal disorders) | 6 (19) | 16 (48)
Weight loss (Investigations) | 6 (12) | 5 (18)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
White blood cell decreased (Investigations) | 31 (122) | 42 (237)
Wound infection (Infections and infestations) | 2 (5) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT01978184/Prot_SAP_000.pdf